CLINICAL TRIAL: NCT04628481
Title: Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess Effect and Safety of 400 mg Twice a Day Oral Ladarixin in Patients With Recent Onset Type 1 Diabetes and Low Residual β-cell Function at Baseline (GLADIATOR)
Brief Title: A Study of Oral Ladarixin in Recent Onset Type 1 Diabetes and a Low Residual β-cell Function
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped due to futility as per protocol
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LDX0319; 2020-001926-71 (EudraCT Number)
Record Dates: First submitted 2020-11-09; First posted 2020-11-13 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Recent Onset type1 Diabetes
Keywords: type1 diabetes
MeSH Terms: interventions — 2'-((4'-trifluoromethanesulfonyloxy)phenyl)-N-methanesulfonylpropionamide; Interleukin-8; Receptors, Interleukin-8B

STUDY DESIGN:
Intervention Model Description: Patients were randomly (2:1) assigned to receive either ladarixin treatment (400 mg b.i.d. for 13 cycles of 14 days on/14 days off - treatment group) or matched placebo (control group). The two groups were balanced within centers.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study proceeded under double-blind condition up to month 18 visit of the last patient randomized. Thereafter, the blind was broken and remaining follow-up will proceeded in an open fashion. This approach allowed to anticipate access to efficacy data without significantly affecting data integrity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ladarixin (Experimental): 400 mg b.i.d. for 13 cycles of 14 days on/14 days off
  Interventions: Drug: Ladarixin
- Placebo (Placebo Comparator): matching placebo b.i.d. for 13 cycles of 14 days on/14 days off
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ladarixin — Oral ladarixin twice a day for 13 cycles
  Other Names: allosteric inhibitor of CXCL8 (IL-8), CXCR1 and CXCR2 receptors
  Arms: Ladarixin
Drug: Placebo — Oral placebo twice a day for 13 cycles
  Arms: Placebo

SUMMARY:
Objectives The objective of this clinical trial is to assess whether ladarixin treatment has an effect to preserve β-cell function and delay the progression of T1D in adolescent and adult patients.

The safety of ladarixin in the specific clinical setting will be also evaluated.

DETAILED DESCRIPTION:
The study will be a phase 2, multicenter, double-blind, placebo-controlled study. It will randomize approximately 130-140 patients (with up to an estimated 15-20% adolescents), with recent onset (within 180 days from 1st insulin administration) type 1 diabetes (T1D), assigned (2:1) to receive either oral ladarixin treatment (400 mg b.i.d. for 13 cycles of 14 days on/14 days off - treatment group) or placebo (control group). Recruitment will be competitive among the study sites, until the planned number of patients is randomized.

Ladarixin and placebo will be both administered for 1 year. All patients will be followed-up for 24 months from the 1st administration of the study medication. After the initial 12-m treatment period, all patients will enter into a 12-month follow-up (total period 24-month after first IMP administration). The study database (DB) will be locked when the last randomized patient has completed the month 12 visit (or being lost in follow-up), and relative data have been fully reconciled and cleaned; at that point, the DB will be unblinded and all endpoints, including the 6-month primary endpoint, will be analyzed, and the follow-up will continue under open-label conditions up to month 24.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 14-45 years, inclusive;
2. Recent onset T1D (1st IMP dose within 180 days from 1st insulin administration);
3. Positive for at least one diabetes-related auto-antibody (anti-GAD; IAA, if obtained within 10 days of the onset of insulin therapy; IA-2 antibody; ZnT8);
4. Require, or has required at some time, insulin therapy through one or more separate subcutaneous injections or Continuous Subcutaneous Insulin Infusion (CSII).
5. Fasting C peptide < 0.205nmol/L;
6. Residual beta-cell function as per peak stimulated (MMTT) C-peptide level >0.2nmol/L; MMTT should not be performed within one week of resolution of a diabetic ketoacidosis event;
7. Patient able to comply with all protocol procedures for the duration of the study, including scheduled follow-up visits and examinations;
8. Patients who have given written informed consent prior of any study-related procedure not part of standard medical care (participants under the age of 18, shall provide an assent for the study as per country requirements). Specific consent must be given by adolescents to be selected for the full PK analysis.

Exclusion Criteria:

1. A type 2 diabetes diagnosis or any other unstable chronic disease for which dose adjustment of specific medication is anticipated during the trial;
2. Moderate to severe renal impairment as per estimated Glomerular Filtration Rate (eGFR) 60 mL/min/1.73m2, as determined using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation;
3. Hepatic dysfunction defined by increased ALT/AST > 3 x upper limit of normal (ULN) and increased total bilirubin > 3 mg/dL [>51.3 μmol/L];
4. Hypoalbuminemia defined as serum albumin < 3 g/dL;
5. QTcF > 470 msec;
6. Occurrence of an episode of ketoacidosis or hypoglycemic coma in the past 2 weeks;
7. A history of significant cardiovascular disease/abnormality;
8. Known hypersensitivity to non-steroidal anti-inflammatory drugs;
9. Concomitant treatment with drugs metabolized by CYP2C9 with a narrow therapeutic index [i.e. phenytoin, warfarin, sulphonylurea hypoglycemics (e.g. tolbutamide, glipizide, glibenclamide/glyburide, glimepiride, nateglinide) and high dose amitriptyline (> 50 mg/day)];
10. Previous (past 2 weeks) and concomitant treatment with antidiabetic agents as metformin, sulfonylureas, glinides, thiazolidinediones, exenatide, liraglutide, DPP-IV inhibitors, SGLT2-inhibitors or amylin, or any medications known to influence glucose tolerance (e.g. beta-blockers, angiotensin-converting enzyme inhibitors, interferons, quinidine antimalarial drugs, lithium, niacin, etc.);
11. Past (past month) or current administration of any immunosuppressive medications (including oral or systemic corticosteroids) and use of any investigational agents, including any agents that impact the immune response or the cytokine system;
12. Significant systemic infection during the 4 weeks before the 1st dose of the study drug (e.g., infection requiring hospitalization, major surgery, or IV antibiotics to resolve; other infections, e.g., bronchitis, sinusitis, localized cellulitis, candidiasis, or urinary tract infections, must be assessed on a case-by-case basis by the investigator regarding whether they are serious enough to warrant exclusion);
13. History of positive status for hepatitis A (IgM), hepatitis B (not due to immunization), hepatitis C and HIV..
14. Pregnant or breast-feeding women. Unwillingness to use effective contraceptive measures up to 2 months after the end of study drug administration (females and males). Effective contraceptive measures include a hormonal birth control (e.g. oral pills, long term injections, vaginal ring, patch); the intrauterine device (IUD); a double barrier method (e.g. condom or diaphragm plus spermicide foam); abstinence.

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 141 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 2-hour AUC of C-peptide response to the Mixed Model Tolerance Test (MMTT) | Month 6
  C-peptide level is an indirect measure of pancreatic beta-cell function. The MMTT was performed after an overnight fast, at baseline

SECONDARY OUTCOMES:
Change from baseline in 2-hour AUC of C-peptide response to the MMTT | Months 12, 18 and 24
Change in HbA1c from baseline | Months 6, 12, 18 and 24
Time in range (TIR) by Continuous Glucose Monitoring (CGM) | Months 6, 12, 18, 24
Proportion of patients with HbA1c <7% who did not experience severe hypoglycemic events during treatment | Months 6, 12, 18, 24
Average (previous 3 days) daily insulin requirement (IU/kg/day) | Months 6, 12, 18, 24
Proportion of patients with HbA1c <7% and daily insulin requirement <0.5 (IU/kg/day) | Months 6, 12, 18, 24
Additional Glucose Variability Indices derived from CGM | Months 6, 12, 18 and 24
  Additional Glucose Variability Indices derived from CGM (glucose AUC outside the target range of 70 - 180 mg/dL, 2-hour postprandial glucose (PPG)).
Additional Glucose Variability Indices derived from MAGE | Months 6, 12, 18 and 24
  Additional Glucose Variability Indices derived from Mean Amplitude Glycemic Excursions (MAGE)
Additional Glucose Variability Indices derived from CONGA-n | Months 6, 12, 18 and 24
  Additional Glucose Variability Indices derived from continuous overall net glycemic action (CONGA)-n
Additional Glucose Variability Indices derived from MODD | Months 6, 12, 18 and 24
  Additional Glucose Variability Indices derived from Mean Of the Daily Differences (MODD).
Additional Glucose Variability Indices derived from mean daily blood glucose, SD | Months 6, 12, 18 and 24
  Additional Glucose Variability Indices derived from mean daily blood glucose, SD (Standard Deviation).
Number of self-reported episodes of severe hypoglycemia | Months 6, 12, 18, 24
  For the purpose of this study, a severe hypoglycemic event is defined as an event with one of the following symptoms: "memory loss, confusion, uncontrollable behavior, irrational behavior, unusual difficulty in awakening, suspected seizure, seizure, loss of consciousness, or visual symptoms", in which the subject was unable to treat him/herself and which was associated with either a blood glucose level <54mg/dL or prompt recovery after oral carbohydrate, i.e. glucose, or glucagon administration.
Percentage of patients not requiring insulin therapy | Months 6, 12, 18, 24
  This outcome aims to assess the % of patients who do not require an insulin therapy
Estimated Glucose Disposal Rate (eGDR) | Months 6, 12, 18, 24
  Estimated Glucose Disposal Rate (eGDR) is a marker for the Assessment of Insulin Resistance and a validated clinical tool for estimating insulin sensitivity in type 1 diabetes.

CONTACTS AND LOCATIONS:
Locations (56):
- United States (25):
  - University of Alabama at Birmingham (UAB) - The Kirklin Clinic (TKC) - Multidisciplinary Comprehensive Diabetes Clinic (MCDC), Birmingham, Alabama
  - Phoenician Centers for Research and Innovation, Phoenix, Arizona
  - University of California San Diego, La Jolla, California
  - Center of Excellence in Diabetes & Endocrinology (CEDE), Sacramento, California
  - University of Colorado School of Medicine - Barbara Davis Center for Childhood Diabetes (BDC) - Specialty Clinic, Aurora, Colorado
  - Christiana Care Endocrinology Specialists, Newark, Delaware
  - Diabetes Care Center - Hudson, Hudson, Florida
  - Global Life Research Network, Miami, Florida
  - AdventHealth (Florida Hospital) - Diabetes Institute - Orlando, Orlando, Florida
  - Atlanta Diabetes Associates (ADA), Atlanta, Georgia
  - The University of Chicago, Chicago, Illinois
  - Prairie Education and Research Cooperative d/b/a Central Illinois Diabetes and Clinical, Springfield, Illinois
  - Indiana University - Riley Hospital for Children, Indianapolis, Indiana
  - The Cotton-O'Neil Diabetes and Endocrinology Center, Topeka, Kansas
  - University of Louisville, Louisville, Kentucky
  - Joslin Diabetes Center, Harvard Medical School, Boston, Massachusetts
  - UBMD Physicians Group - Pediatrics - Conventus, Buffalo, New York
  - "WakeMed Physician Practices - Pediatric Endocrinology - WakeMed Raleigh Medical Park Location", Raleigh, North Carolina
  - University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Pittsburgh - UPMC, Pittsburgh, Pennsylvania
  - Cook Children's Endocrinology and Diabetes Program, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - Eastern Virginia Medical School (EVMS) - Strelitz Diabetes Center, Norfolk, Virginia
- Belgium (3):
  - Clinique du Sud Luxembourg - Vivialia-Arlon, Arlon
  - Universitair Ziekenhuis Brussel (UZB), Jette
  - General Hospital AZ Nikolaas, Sint-Niklaas
- Georgia (4):
  - Aleksandre Aladashvili Clinic LLC, Tbilisi
  - National Center for Diabetes Research LTD, Tbilisi
  - National Institute of Endocrinology LTD, Tbilisi
  - Tbilisi Heart and Vascular Clinic LTD, Tbilisi
- Germany (6):
  - Medical Center - University of Freiburg, Freiburg im Breisgau
  - Universitaetsklinikum Gessen und Marburg GmbH - Medizinische Klinik und Poliklinik III, Glessen
  - Diabestesinstitut Heidelberg, Heidelberg
  - Die Praxis am Ludwigsplatz, Ludwigshafen am Rhein
  - Institut fuer Diabetes forschung in Muenster (IDFM), Münster
  - Schwerpunktpraxis fuer Diabetes & Ernaehrungsmedizin, Münster
- Israel (3):
  - Soroka Medical Center, Beersheba
  - Schneider Children's Medical Center, Petah Tikva, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (10):
  - Ospedale Pediatrico G. Salesi - Centro Regionale di Diabetologia Clinica Pediatrica, Ancona
  - Azienda Ospedaliero-Universitaria Conzorziale Policlinico di Bari, Bari
  - Università degli Studi Magna Graecia di Catanzaro, Azienda Ospedaliero-Universitaria Mater Domini, Catanzaro
  - Universitá degli Studi di Milano - Ospedale Luigi Saco, Milan
  - Centro regionale di Diabetologia Pediatrica "G. Stoppoloni", Azienda Ospedaliera Universitaria "Luigi Vanvitelli", Napoli
  - Azienda Ospedaliera Universitaria Policlinico "Paolo Giaccone", Palermo
  - Università Campus Bio-Medico di Roma (UCBM) - Policlinico Universitario, Roma
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale Pediatrico Bambino Gesu, Roma
  - Universita Cattolica del Sacro Cuore - Policlinico Universitario "Agostino Gemelli", Roma
  - "Sapienza" Università di Roma- Azienda Ospedaliero Universitaria Policlinico Umberto I, Rome
- Serbia (4):
  - Clinical Center of Serbia, Clinic for Endocrinology, Diabetes and Metabolic Diseases, Belgrade
  - University Children's Hospital, Belgrade
  - Clinical center Kragujevac, Clinic for internal diseases, Center for endocrinology, diabetes and metabolic diseases, Kragujevac
  - Clinical Center Nis, Clinic for endocrinology, Niš
- University Children's Hospital, University Medical Center Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No